CLINICAL TRIAL: NCT01447745
Title: Visceral Obesity/Ectopic Fat and Non-invasive Markers of Atherosclerosis: A Cardiometabolic-cardiovascular Imaging Study
Brief Title: Abdominal Fat and Imaging Measurements of Heart Disease
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jean-Pierre DESPRÉS, PhD, Principal Investigator, Laval University
Other Study IDs: CIHR MOP-114920
Record Dates: First submitted 2011-09-27; First posted 2011-10-06 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Visceral Obesity; Atherosclerosis; Metabolic Syndrome
Keywords: Visceral obesity; Cardiometabolic risk; Atherosclerosis; Ectopic fat; Carotid plaque; Magnetic resonance imaging (MRI); Computed tomography (CT)
MeSH Terms: conditions — Obesity, Abdominal; Atherosclerosis; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, white cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational, longitudinal study: Adult men and women representative of the population of asymptomatic adult men and women aged from 35-65 years living in the Québec City metropolitan area

SUMMARY:
Although it is frequently mentioned in the media that overweight and obesity have reached epidemic proportions worldwide and in this country, some Canadians are perplexed and sometimes confused about the role of obesity in diabetes and heart disease. In fact, the investigators even hear from time to time that there could be "healthy" obese individuals. In clinical practice, assessment of obesity as a risk factor for cardiovascular disease (CVD) remains a challenge as even some physicians are confused. However, studies conducted in our laboratory and by other research teams around the world over the last 20 years have clearly shown that body shape is more important than body size when evaluating the risk of overweight/obesity and that high accumulation of abdominal fat (excess belly fat) increases the risk of diabetes and cardiovascular disease (CVD).

The investigators now need to better understand the link between excess belly fat and atherosclerosis (the thickening of artery walls by fatty deposits, also referred to as atherosclerotic plaque), leading to complications such as angina (chest pain) and myocardial infarction (heart attacks). Using non-invasive imaging techniques such as magnetic resonance imaging, the investigators therefore propose to examine the relationships between measures of fatness and of abdominal fat and the size of atherosclerotic plaque in large blood vessels of apparently healthy human subjects. This study is also a unique opportunity to look, for the first time, at the relationship between belly fat, blood sugar, several well-known risk factors for heart disease (cholesterol, blood pressure, cardiorespiratory fitness, etc.) and the size of atherosclerotic plaques. This research program should pave the way to the development of new improved preventive/therapeutic approaches focusing not on body weight but rather on abdominal fat and associated blood abnormalities which are predictive of the development of atherosclerotic plaques leading to the premature development of heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 35-65 years

Exclusion Criteria:

* Massive obesity (BMI ≥ 40 kg/m2)
* Pharmacological treatment for lipids, hypertension and/or type 2 diabetes
* Clinical signs of cardiovascular disease
* Chronic inflammatory or auto-immune diseases
* Pulmonary diseases on corticosteroids
* Cancers not in remission
* History or clinical evidence of coronary heart disease (CHD)
* History of revascularisation procedures
* Current smoking
* Hormonal replacement therapy

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random sample of adult men and women representative of the population of asymptomatic adult men and women aged from 35-65 years living in the Québec City metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 357 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Change in carotid vessel wall volume measured by magnetic resonance imaging (MRI) | Change between baseline and 3-year follow-up
  Cross-sectional and longitudinal analyses of the relationships between indices of body fat distribution, visceral adiposity/ectopic fat deposition, cardiorespiratory fitness and non-invasive measurements of macrovascular atherosclerosis

SECONDARY OUTCOMES:
Change in abdominal adipose tissue measured by computed tomography (CT) | Change between baseline and 3-year follow-up
  Visceral and subcutaneous adipose tissue will be determined at both L2-L3 and L4-L5 levels
Change in epi- and pericardial fat measured by magnetic resonance imaging (MRI) | Change between baseline and 3-year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: DESPRÉS Jean-Pierre, PhD, Principal Investigator — Université Laval/Institut universitaire de cardiologie et de pneumologie de Québec
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Canada